CLINICAL TRIAL: NCT05887024
Title: Effect of Shock Wave Therapy on Low Back Pain and Sciatica in Patients With Post-laminectomy Fibrosis
Brief Title: Effect of Shockwave Therapy on Post-laminectomy Fibrosis Low Back Pain Patients.
Acronym: SWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marwa Mohamed Hany Sedeek Abousenna (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Hany Sedeek Abousenna, physiotherapist Marwa Mohamed Hany Sedeek Abousenna, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004382
Record Dates: First submitted 2023-04-28; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Post-laminectomy Syndrome
Keywords: Sciatica; low back pain; post-laminectomy syndrome; Radial Shock Wave Therapy
MeSH Terms: conditions — post laminectomy syndrome; Sciatica; Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: A. Control group (Group A) thirty patients will receive conventional physical therapy program (TENS, electric heating packs, and McKenzie back exercises).
  B. Study group (Group B) thirty patients will receive radial extracorporeal shock wave therapy and conventional physical therapy program (TENS, electric heating packs, and McKenzie back exercises).
Who Masked: Participant
Masking Description: The selected patients will be allocated by computerized block randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled (Other): thirty patients will receive conventional physical therapy program (TENS, electric heating packs, and McKenzie back exercises).
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Procedure: McKenzie Back exercises; Device: electric heating pads
- shock wave therapy (Active Comparator): thirty patients will receive radial extracorporeal shock wave therapy and conventional physical therapy program (TENS, electric heating packs, and McKenzie back exercises).
  Interventions: Device: Radial Extracorporeal Shock wave Therapy; Device: Transcutaneous Electrical Nerve Stimulation (TENS); Procedure: McKenzie Back exercises; Device: electric heating pads

INTERVENTIONS:
Device: Radial Extracorporeal Shock wave Therapy — Shock wave therapy: (BECO) S/N 16B011375
  Arms: shock wave therapy
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — EME (Therapic 9400) TENS
Procedure: McKenzie Back exercises — Graduated Progressive back exercise program.
Device: electric heating pads — electrical conducting heat pack.

SUMMARY:
The aim of this study is clinical trial to investigate the effect of Radial Extracorporeal Shock wave therapy in patients with sciatica and low back pain caused by post laminectomy scarring. the study will answer the following question:

1. what is the effect of Shock Wave Therapy on low back pain and sciatica caused by post-laminectomy fibrosis? patients in the study group will receive radial extracorporeal shock wave therapy and conventional physical therapy program (TENS, electric heating packs, and McKenzie back exercises).

ELIGIBILITY:
Inclusion Criteria:

1. Recruited patients will be diagnosed by neurosurgeon as sciatic pain and low back pain caused by post laminectomy scarring.
2. Both genders will be recruited.
3. Their age will range from: 30-50 years (Sharaf, et al., 2022).
4. Recruited patients will be randomly assigned in to two equal groups.
5. Unilateral radicular sciatica.
6. Constant back pain OR aggravated by movement,
7. Restricted lumbar range of motion.
8. Tenderness at the site of incision.
9. Duration of symptoms: three weeks to six months postoperatively

Exclusion Criteria:

1. Past history of vertebral fracture.
2. Spinal cord compression.
3. Vertebral tuberculosis.
4. Polyneuropathy.
5. Diabetic peripheral neuropathy.
6. Spinal tumor.
7. Recurrent disc herniation after surgery.
8. Spondylolisthesis.
9. Vascular diseases, e.g., peripheral vascular diseases, coronary artery bypass graft and coagulation diseases.
10. Potential pregnancy.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 4 weeks
  The VAS consisted of a 10 cm horizontal line with the description "no pain" on the far left and "worst possible pain" on the far right

SECONDARY OUTCOMES:
Pain algometry | 4 weeks
  PainTest™ FPX 25 Algometer (Wagner Instruments, Greenwich, USA)
Lumbar Range Of Motion | 4 weeks
  The BROM II
The Oswestry Disability Index: (ODI) | 4 weeks
  The Oswestry disability index is a self-completed, valid tool with adequate reliability to identify changes in functional disability
Sensory Nerve Conduction Study (NCS) | 4 weeks
  Sensory nerve action potentials (sensory nerve amplitude)

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be free to share within 6 months to 1 year after publication.
Supporting Information: Study Protocol
Time Frame: 6 months to 1 year after publication.